CLINICAL TRIAL: NCT03013504
Title: A Randomised, Double-blind, Parallel Group, Equivalence, Multicentre Phase III Trial to Compare the Efficacy, Safety and Pharmacokinetics of HD201 to Herceptin® in Patients with HER2+ Early Breast Cancer
Brief Title: A Phase III Trial to Compare the Efficacy, Safety and Pharmacokinetics of HD201 to Herceptin® in HER2+ Early Breast Cancer Patients
Acronym: TROIKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prestige Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TROIKA
Record Dates: First submitted 2016-12-29; First posted 2017-01-06 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2023-02

CONDITIONS: HER2 Positive Breast Cancer
Keywords: randomized; double-blind; parallel group; equivalence; multicentre; phase III; efficacy; safety; pharmacokinetics; HD201; docetaxel; Herceptin; HER2 positive; breast cancer; early breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Docetaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HD201 in combination with docetaxel (Experimental): 8 mg/kg i.v. loading dose over 90 mins in Cycle 1 and 6 mg/kg i.v. dose every 3 weeks over 60 mins then 30 mins for subsequent cycles (cycles 2-8), followed by surgery, then adjuvant period of 8mg/kg i.v. loading dose over 90 mins in cycle 9, and subsequent 6mg/kg (if therapy is missed by >1 week, a re-loading dose of 8mg/kg should be given) over 30 mins for subsequent 9 cycles (cycles 10-18), disease progression, unacceptable toxicity, non-compliance, or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever occurs first.
  Neoadjuvant chemotherapy:
  Cycles 1-4: Docetaxel 75 mg/m² on day 1 of each 3-weeks cycle via 1h i.v. Infusion Cycles 5-8: EC on day 1 of each 3-weeks cycle: Epirubicin 75 mg/m² via 3-30 mins i.v. Infusion, Cyclophosphamide 500 mg/m² via 3-30 mins i.v. Infusion
  Interventions: Drug: HD201; Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide
- Herceptin® in combination with docetaxel (Active Comparator): 8 mg/kg i.v. loading dose over 90 mins in Cycle 1 and 6 mg/kg i.v. dose every 3 weeks over 60 mins then 30 mins for subsequent cycles (cycles 2 -8) for cycles 2-8, followed by surgery, and subsequent adjuvant period of 8mg/kg i.v. loading dose over 90 mins in cycle 9, then 6mg/kg (if therapy is missed by >1 week, a re-loading dose of 8mg/kg should be given) over 30 mins for subsequent 9 cycles (cycles 10-18), disease progression, unacceptable toxicity, non-compliance, or withdrawal of consent by the patient, or the investigator decides to discontinue treatment, whichever occurs first.
  Neoadjuvant chemotherapy:
  Cycles 1-4: Docetaxel 75 mg/m² on day 1 of each 3-weeks cycle via 1h i.v. Infusion Cycles 5-8: EC on day 1 of each 3-weeks cycle: Epirubicin 75 mg/m² via 3-30 mins i.v. Infusion, Cyclophosphamide 500 mg/m² via 3-30 mins i.v. Infusion
  Interventions: Drug: Herceptin; Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: HD201 — Loading dose of 8mg/kg in Cycle 1 and 6mg/kg in subsequent cycles.
  Other Names: Trastuzumab
  Arms: HD201 in combination with docetaxel
Drug: Herceptin — Loading dose of 8mg/kg in Cycle 1 and 6mg/kg in subsequent cycles.
  Other Names: Trastuzumab
  Arms: Herceptin® in combination with docetaxel
Drug: Docetaxel — 75mg/m2 via i.v. infusion during cycles 1 to 4.
Drug: Epirubicin — 75 mg/m2 via i.v. infusion during cycles 5-8.
Drug: Cyclophosphamide — 500 mg/m2 via i.v. infusion during cycles 5-8.

SUMMARY:
In the TROIKA study, the proposed biosimilar HD201 will be compared to its reference product Herceptin®. The aim of the study is to demonstrate equivalence of HD201 and Herceptin® in terms of efficacy, safety and pharmacokinetics.

DETAILED DESCRIPTION:
This is a randomised, double-blind, parallel group, equivalence, multicentre Phase III study. 500 patients with HER2+ early breast cancer (EBC) will be randomised (1:1) to receive either HD201 in combination with chemotherapy (n=250) or Herceptin® in combination with chemotherapy (n=250).

HD201 or Herceptin® will be administered every 3 weeks for 8 cycles(24 weeks). After administration of the final neoadjuvant study drug dose, surgery will be done within 3-8 weeks followed by an adjuvant treatment period for 10 cycles.

Patients completing the 18 cycles of treatment and those discontinuing the study will attend an End of Treatment (EOT) visit 4 weeks (+/- 2 days), after last administration of study medication, followed by a follow-up period of 2 years.

Patients will attend study visits every 3 weeks. At each visit, patients will undergo a complete physical examination, vital signs, weight, performance status, clinical laboratory tests and adverse events (AEs), concomitant medication will be recorded. After the EOT visit patients will be followed every 6 months for an additional 24 months or until death, whichever occurs first, to collect data on cardiac safety and disease status.

Cardiac safety will be assessed by echocardiography or multigated acquisition (MUGA) scan to evaluate the left ventricular ejection fraction (LVEF) (at screening, before cycle 5, before surgery, before cycles 12 and 16, EOT visit, and at 6 and 12 months after the completion of trastuzumab (more frequent if necessary)) and by means of a 12-lead ECG (at screening, before cycle 5, before surgery, before cycles 12 and 16, EOT visit, and at 6 and 12 months after the completion of trastuzumab).

The primary efficacy endpoint, total pathological complete response (tpCR) will be assessed at the time of surgery after neoadjuvant treatment completion after 24 weeks. tpCR will be assessed both by local and by central reading.

Sampling for pharmacokinetics (PK) analysis (determination of Ctrough values) will be performed in all patients before cycle 5 and cycle 8.

An Independent Data Monitoring Committee will be implemented that reviews accumulating data of the clinical trial with respect to any potential safety issues, study progress and critical efficacy endpoints. The members will be selected on the basis of relevant experience and understanding of clinical research and the issues specific to the therapeutic area, as well as previous data monitoring committee experience.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Females ≥ 18 years of Age
3. Eastern Cooperative Oncology Group (ECOG) performance Status (PS) < 2.
4. Known Hormone receptor (oestrogen receptor and progesterone receptor) status.
5. HER2 overexpressed as assessed by

   1. Immunohistochemistry (IHC) or
   2. Fluorescent in situ hybridisation (FISH); FISH positive is defined as FISH amplification Ratio ≥ 2.0 / number of HER2 gene copies per cell >2
   3. Chromogenetic in stu hybridisation (CISH) positive
   4. Patients with IHC score 3+ or positive FISH/CISH test
   5. Patients with an IHC score 2+ must also have a positive FISH/CISH test
6. LVEF ≥ 50% or within the normal Level of the Institution, as assessed by echocardiography or MUGA scan.
7. Life expectancy > 12 weeks.
8. Adequate bone marrow function as evidenced by the following:

   1. Absolute neutrophils count ≥ 1,500/μL
   2. Haemoglobin ≥ 9 g/dL
   3. Platelet count ≥ 100,000/μL Up to 5% Deviation is acceptable.
9. Adequate hepatic and renal function as evidenced by the following:

   1. Creatinine clearance ≥ 60mL/min
   2. total Bilirubin ≤ 1.5x upper limit of normal (ULN)
   3. AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN Up to 10% deviation is acceptable.
10. Ability to comply with the study protocol.
11. Female patients of childbearing potential must have a negative Serum pregnancy test within 7 days prior to first dose of study treatment and agree to use effective contraception (intrauterine device, diaphragm, diaphragm with spermicide or a reliable barrier method, eg condom with spermicide) throughout the study period and 7 months after discontinuation of study drug.
12. Non-metastatic, unilateral, newly diagnosed, operable early breast cancer (EBC) of clinical stage II and III including inflammatory breast cancer. Histologically confirmed primary invasive carcinoma of the breast.

Exclusion Criteria:

Patients meeting any of the following criteria must not be enrolled in the study:

1. Metastatic (stage IV) with exception of supraclavicular nodes.
2. Bilateral breast cancer
3. Multicentric breast cancer
4. History of any prior invasive breast carcinoma, except for subjects with a past history of ductal carcinoma in situ (DCIS) treated with surgery.
5. History of malignant neoplasms within 5 years prior to randomisation, except for curatively treated carcinoma in situ of uterine cervix, basal cell carcinoma of the skin or squamous cell carcinoma of the skin (malignant neoplasms occurring more than 5 years prior to randomisation are permitted if curatively treated with surgery only).
6. Previous history of radiation therapy, anti-neoplastic immunotherapy, chemotherapy or anti-neoplastic biotherapy (including prior HER2 directed therapy).
7. Major surgery within 2 weeks prior to randomisation
8. Serious cardiac illness that would preclude the use of trastuzumab such as:

   * history of documented congestive heart failure (CHF) (New York Heart Association, NYHA, class III or greater heart disease)
   * LVEF < 50% by echocardiography or MUGA scan
   * angina pectoris requiring anti-anginal medication
   * evidence of transmural infarction on electrocardiogram (ECG)
   * uncontrolled hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg)
   * clinically significant valvular heart disease
   * high-risk uncontrolled arrhythmias.
9. Serious pulmonary illness enough to cause dyspnoea at rest or requiring supplementary oxygen therapy.
10. Known history of active hepatitis B virus (HBV) and active hepatitis C virus (HCV) infection.
11. Known HIV infection by patient declaration.
12. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
13. Known hypersensitivity to the IMPs, non-IMPs or any of the ingredients or excipients of the IMPs or non-IMPs.
14. Known hypersensitivity to murine proteins.
15. Pre-existing peripheral sensory or motor neuropathy ≥ grade 2 (as defined by NCI-CTCAE v4.03).
16. Lactating or pregnant woman. A pregnancy test is required for all women of childbearing potential including women who had menopause onset within 2 years prior to randomisation. Women of childbearing potential must agree to use contraceptive methods during the study and for 7 months after the last dose of IMP.
17. Participation in any clinical study or having taken any investigational therapy during the 1-month period immediately preceding administration of the first dose.
18. Patients unwilling to follow the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
total pathological complete response rate (tpCR) | After 24 weeks (end of cycle 8)
  To compare the total pathological complete response rate (tpCR) in patients treated with HD201 plus chemotherapy to that in patients treated with Herceptin® plus chemotherapy.

SECONDARY OUTCOMES:
total breast pathological complete response rate (bpCR) | After 24 weeks (end of cycle 8)
  To compare total breast pathological complete response rate (bpCR) between the two arms at the time of surgery.
Overall response rate (ORR) | After 24 weeks (end of cycle 8)
  ORR defined as proportion of patients whose best overall response is either complete response (CR) or partial response (PR) at the time of surgery.
Overall Survival (OS) | From date of randomisation until death from any cause or two years after End of Treatment, whichever comes first
  OS defined as the time from Day 1 of therapy until death from any cause
Event-free Survival (EFS) | From date of randomisation until death from any cause or two years after End of Treatment, whichever comes first
  EFS defined as the time from Day 1 of therapy (day of first infusion of medication on study) until progression of disease or death from any cause.
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | From baseline through study completion until 18 months or until death, whichever came first
  Safety and tolerability will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events and CTC v4.03
Cardiac dysfunction | Within 28 days before start of treatment, before cycle 5,12 and 16 (1 cycle is 3 weeks), before surgery (after 24 weeks), at end of treatment (4 weeks from last administration of drug medication) and one year after completion of trastuzumab therapy.
  Cardiac dysfunction will be monitored by 12-Lead ECG and measurement of the LVEF by echocardiography or MUGA scan
Immunogenecity | At baseline (within 28 days before start of treatment), before surgery (after 24 weeks), at end of treatment (4 weeks from last administration of drug medication) and one year after completion of trastuzumab therapy.
  Incidence of human trastuzumab antibodies
Clearance (Pharmacokinetic) | Before administration of treatment at Cycles 5 and 8 (1 cycle is 3 weeks)
  Sampling will be performed in all patients to compare the PK through values of HD201 and Herceptin.
Area under the curve (AUC, Pharmacokinetic) | Before administration of treatment at Cycles 5 and 8 (1 cycle is 3 weeks)
  Sampling will be performed in all patients to compare the PK through values of HD201 and Herceptin.
Plasma half life (Pharmacokinetic) | Before administration of treatment at Cycles 5 and 8 (1 cycle is 3 weeks)
  Sampling will be performed in all patients to compare the PK through values of HD201 and Herceptin.

CONTACTS AND LOCATIONS:
Locations (15):
- Minsk Clinical Oncological Dispensary, Minsk, Belarus
- Complex Oncology Center, Plovdiv, Bulgaria
- East Tallinn Central Hospital, Tallinn, Estonia
- Centre René Huguenin (Institut Curie), Saint-Cloud, France
- S. Khechinashvili University Hospital, Tbilisi, Georgia
- Hungary (2):
  - National Institute of Oncology, Budapest
  - University of Debrecen, Debrecen
- Modena Hospital, Modena, Italy
- Malaysia (2):
  - Beacon International Specialist Centre, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur
- Szpital Specjalistyczny Brzeziny, Brzeziny, Poland
- LLC "Vitamed", Moscow, Russia
- Hospital Universitario Virgen Macarena, Seville, Spain
- Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Thailand
- GI "V. T. Zaycev Institute General and Urgent Surgery of NAMS of Ukraine ", Kharkiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivot X, Manikhas AG, Shamrai V, Dzagnidze G, Soo Hoo HF, Kaewkangsadan V, Petrelli F, Villanueva C, Kim J, Pradhan S, Jaison L, Feyaerts P, Kaufman L, Derde MP, Deforce F, Cox DG. Final analysis of the phase 3 randomized clinical trial comparing HD201 vs. referent trastuzumab in patients with ERBB2-positive breast cancer treated in the neoadjuvant setting. BMC Cancer. 2023 Jan 31;23(1):112. doi: 10.1186/s12885-023-10574-2. PMID 36721174
- [Derived] Pivot X, Georgievich MA, Shamrai V, Dzagnidze G, Soo Hoo HF, Kaewkangsadan V, Petrelli F, Villanueva C, Nikolaevich LO, Hii J, Kim J, Pradhan S, Jaison L, Feyaerts P, Kaufman L, Derde MP, Bonamy GMC, Deforce F, Cox DG. Efficacy of HD201 vs Referent Trastuzumab in Patients With ERBB2-Positive Breast Cancer Treated in the Neoadjuvant Setting: A Multicenter Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 May 1;8(5):698-705. doi: 10.1001/jamaoncol.2021.8171. PMID 35238873